CLINICAL TRIAL: NCT06306755
Title: Effectiveness of Risk-based Sequential Screening for Esophageal and Gastric Cancer: A Community-Based Randomized Controlled Trial
Brief Title: Effectiveness of Risk-based Sequential Screening for Esophageal and Gastric Cancer
Acronym: ERSS-EGC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2021YFC2500405
Record Dates: First submitted 2024-03-03; First posted 2024-03-12 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Cancer; Gastric Cancer; Precision Screening; Sequential Screening; Risk Stratification
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Risk Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequential screening group (Experimental): The enrolled participants will undergo a questionnaire investigation and receive a risk assessment for esophageal and gastric malignancies based on two questionnaire-based diagnostic models. Participants identified as "high-risk" (i.e., with a top 50% risk level) for esophageal and/or gastric malignancy will receive the standard upper gastrointestinal endoscopy. Standardized diagnosis and treatment recommendations will be provided to patients with screening-detected malignant lesions, and green referral channels will be established for them. For participants with screening-detected premalignant lesions, the risk of progression will be evaluated based on endoscopic characteristics, pathological diagnosis, and biomarkers. Individualized reexamination and surveillance will be implemented accordingly.
  Interventions: Procedure: Risk Assessment and Individualized Surveillance
- Universal screening group (Active Comparator): The enrolled participants will undergo a questionnaire investigation and receive the same standard upper gastrointestinal endoscopy as those in the sequential screening group, irrespective of the results of the risk assessment. Standardized diagnosis and treatment recommendations will be provided to patients with screening-detected malignant lesions, and green referral channels will be established for them. For participants with screening-detected premalignant lesions, the reexamination and surveillance will be performed according to the current guidelines for UGIC screening and clinical treatment.
  Interventions: Procedure: Universal screening

INTERVENTIONS:
Procedure: Risk Assessment and Individualized Surveillance — 1. An epidemiological questionnaire-based risk assessment for UGIC conducted prior to the endoscopic examination;
  2. Individuals identified as "high-risk" receive the upper gastrointestinal endoscopic examination with Lugol's Iodine in the esophagus and indigo carmine staining in the stomach;
  3. Individualized reexamination and surveillance strategy will be given to participants diagnosed with premalignant lesions, based on evaluation of risk progression using endoscopic characteristics, pathological diagnosis, and biomarkers.
  Arms: Sequential screening group
Procedure: Universal screening — 1. A questionnaire investigation;
  2. All participants undergo the upper gastrointestinal endoscopic examination with Lugol's Iodine in the esophagus and indigo carmine staining in the stomach;
  3. Reexamination and surveillance will be performed according to the current guidelines for UGIC screening and clinical treatment.
  Arms: Universal screening group

SUMMARY:
To evaluate the feasibility, applicability, effectiveness, and health-economic value of the risk-based sequential screening modality for esophageal and gastric cancers, the investigators aim to initiate a community-based randomized controlled trial in Xun County, Henan Province, which is a high-risk region of upper gastrointestinal cancer (UGIC) in northern China.

A total of 258 target villages from all the 11 communities (townships and streets) in Xun County will be randomly selected and assigned to the sequential screening group and the universal screening group at a ratio of 2:1 and the total sample size will be 21,000.

In the sequential screening group, participants in the top 50% risk level (i.e., stratified as the high-risk subgroup) will be offered a standard upper gastrointestinal endoscopic screening. In contrast, all participants in the universal screening group will receive the endoscopic examination. The surveillance strategy for participants with screening-detected premalignant lesions in the sequential screening group will be tailored based on individualized risk assessment using endoscopic characteristics, pathological diagnosis, and biomarkers. Surveillance for participants in the universal screening group will adhere to current guidelines for UGIC screening and clinical treatment.

Detection rates of upper gastrointestinal malignant lesions, early-stage malignant lesions and premalignant lesions, and health-economic indicators such as the unit cost per detected malignant lesions will be compared between the two groups.

DETAILED DESCRIPTION:
A series of challenges have arisen for the current UGIC screening modality in China, including high screening costs, low detection rates, delayed and unstandardized treatment, and lack of sustainability and scalability. These challenges significantly hinder the normalization and high-quality implementation of UGIC prevention and control efforts. The precision shift in the screening modality is expected to result in substantial savings in medical resources while maximizing the identification and management of high-risk populations.

The investigators aim to initiate a community-based randomized controlled trial to evaluate the effectiveness of risk-stratification-based sequential screening for esophageal and gastric cancer (ERSS-EGC trial) in Xun County of Henan Province, which is a high-risk region of UGIC in northern China.

According to the baseline data obtained from our prior UGIC screening program conducted in the same region, the detection rate of upper gastrointestinal malignant lesions in the targeted population (aged 50-69 years) in the universal screening group is estimated to be 1.1%. It is assumed that the implementation of sequential screening will increase this detection rate by 70%, indicating an expected detection rate of 1.9% for upper gastrointestinal malignant lesions in the sequential screening group. Ultimately, a total of 7,674 endoscopies (with 3,837 in each group) will be required to achieve a statistical power of 80% at a one-sided significance level of 2.5%.

Based on the estimated population coverage determined by sample size, a total of 258 target villages from all the 11 communities (townships and streets) in Xun County will be randomly selected, stratified by townships and streets. These 258 target villages will be randomly assigned to either the sequential screening group or the universal screening group at a ratio of 2:1, based on the population size of each village and stratified by region (urban and rural areas). This results in 172 villages in the sequential screening group and 86 villages in the universal screening group. Approximately 21,000 permanent residents aged 50 to 69 residing in the target villages will be enrolled in the trial.

All enrolled eligible participants will receive an epidemiological questionnaire investigation (collecting data on basic information, dietary habits, environmental exposure, family history, symptoms, quality of life, etc.). Additionally, participants will receive a physical examination, which includes measurement of height, weight, blood pressure, as well as the collection of biological samples. These samples comprise: (1) peripheral venous blood samples for serological screening of infectious diseases, complete blood count, and biospecimen banking (including serum, plasma, white blood cells, and cell-free DNA); (2) tongue coating swab. Furthermore, standardized digital tongue images will be captured from all study participants.

In the sequential screening group, all enrolled participants will be offered a risk assessment for esophageal and gastric malignancies based on two questionnaire-based diagnostic models. Participants identified as "high-risk" (i.e., with a top 50% risk level) for esophageal and/or gastric malignancy will receive the standard upper gastrointestinal endoscopy. Standardized diagnosis and treatment recommendations will be provided to patients with screening-detected malignant lesions, and green referral channels will be established for them. For participants with screening-detected premalignant lesions, the risk of progression will be evaluated based on endoscopic characteristics, pathological diagnosis, and biomarkers. Individualized reexamination and surveillance will be implemented accordingly.

In the universal screening group, all enrolled participants will receive the same standard upper gastrointestinal endoscopy as those in the sequential screening group, irrespective of the results of the risk assessment. Standardized diagnosis and treatment recommendations will be provided to patients with screening-detected malignant lesions, and green referral channels will be established for them. For participants with screening-detected premalignant lesions, the reexamination and surveillance will be performed according to the current guidelines for UGIC screening and clinical treatment.

Prior to the endoscopic examination, exfoliated cells from the esophagus and esophagogastric junction will be collected using a sponge device and stored in preservation solution for subsequent scientific research. For individuals who exhibited abnormalities during endoscopic examination and are biopsied for pathologic diagnosis, a paired tissue biopsy sample at the same location will be collected and preserved in RNA protection solution for further scientific research.

The primary outcome of this study is the detection rate of upper gastrointestinal (esophageal/gastric) malignant lesions. The secondary outcomes include the rate of early-stage upper gastrointestinal (esophageal/gastric) malignant lesions, detection rate of upper gastrointestinal (esophageal/gastric) premalignant lesions, response rate of endoscopic examination, total screening costs, unit cost per detected upper gastrointestinal malignant lesions, unit cost per detected early-stage upper gastrointestinal malignant lesions, unit cost per detected upper gastrointestinal premalignant lesions, satisfaction of project executors and participants, rate of timely treatment, UGIC-specific mortality, all-cause mortality, and quality of life.

Through a comprehensive comparison with the universal screening, this trial will provide high-level evidence regarding the feasibility, applicability, effectiveness, and health-economic value of the sequential screening modality. Furthermore, it could effectively facilitate standardized diagnosis and treatment for screening-detected patients, providing crucial practical experience and scientific evidence for the reform and development of secondary prevention strategies for UGIC in China.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residency in the target villages in Xun County, Henan Province, China;
* Aged 50 to 69 at the enrollment;
* Voluntarily participate in this study and provide informed consent.

Exclusion Criteria:

* Had a history of endoscopic examination within 5 years prior to the initial interview;
* Had a history of cancer;
* Had a history of mental disorder;
* Positive for hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV);
* Had severe cardiovascular and cerebrovascular diseases;
* Had severe respiratory disease, dyspnea, or asthmaticus status;
* Had retropharyngeal abscess, severe spinal deformity, or aortic aneurysm;
* With physical debility unable to tolerate endoscopic examination, or with difficulty in achieving sedation and self-control;
* In the acute phase of corrosive inflammation of the upper gastrointestinal tract, or with suspected perforation of the upper gastrointestinal tract;
* Had massive ascites, severe abdominal distension, or severe esophageal varices;
* Pregnancy;
* Had severe history of allergies;
* Had propensity for bleeding (coagulopathy);
* Others unable to tolerate the clinical examinations involved in this study.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21000 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of upper gastrointestinal (esophageal/gastric) malignant lesions | 12 months
  Number of detected malignant lesions / Number of completed endoscopies × 100%

SECONDARY OUTCOMES:
Rate of early-stage upper gastrointestinal (esophageal/gastric) malignant lesions | 12 months
Detection rate of upper gastrointestinal (esophageal/gastric) premalignant lesions | 12 months
Response rate of endoscopic examination | 12 months
Total screening costs | 12 months
Unit cost per detected upper gastrointestinal (esophageal/gastric) malignant lesions | 12 months
Unit cost per detected early-stage upper gastrointestinal (esophageal/gastric) malignant lesions | 12 months
Unit cost per detected upper gastrointestinal (esophageal/gastric) premalignant lesions | 12 months
Satisfaction with the risk-based sequential screening modality | 12 months
  Satisfaction with the risk-based sequential screening modality is measured through a one-on-one interview using a semi-structured questionnaire specially designed for this trial.
Rate of timely treatment | 12 months
UGIC-specific mortality | 5-10 years
All-cause mortality | 5-10 years
Quality of life Scale Score | 12 months
  European Quality of Life 5-Dimension (EQ-5D) index score is used to assess health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of genetics, Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Zheng H, Liu Z, Chen Y, Ji P, Fang Z, He Y, Guo C, Xiao P, Wang C, Yin W, Li F, Chen X, Liu M, Pan Y, Liu F, Liu Y, He Z, Ke Y. Development and external validation of a quantitative diagnostic model for malignant gastric lesions in clinical opportunistic screening: A multicenter real-world study. Chin Med J (Engl). 2024 Oct 5;137(19):2343-2350. doi: 10.1097/CM9.0000000000002903. Epub 2024 Feb 26. PMID 38403900
- [Background] Liu Z, Zheng H, Liu M, He Y, Chen Y, Ji P, Fang Z, Xiao P, Li F, Guo C, Yin W, Pan Y, He Z, Ke Y. Development and External Validation of an Improved Version of the Diagnostic Model for Opportunistic Screening of Malignant Esophageal Lesions. Cancers (Basel). 2022 Nov 30;14(23):5945. doi: 10.3390/cancers14235945. PMID 36497427
- [Background] He Z, Liu Z, Liu M, Guo C, Xu R, Li F, Liu A, Yang H, Shen L, Wu Q, Duan L, Li X, Zhang C, Pan Y, Cai H, Ke Y. Efficacy of endoscopic screening for esophageal cancer in China (ESECC): design and preliminary results of a population-based randomised controlled trial. Gut. 2019 Feb;68(2):198-206. doi: 10.1136/gutjnl-2017-315520. Epub 2018 Jan 6. PMID 29306867